CLINICAL TRIAL: NCT00432575
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Fixed-Dose, 8-Week Treatment, Multi-Center Trial Evaluating the Efficacy and the Safety of 3 Oral Doses of Surinabant as an Aid to Smoking Cessation in Cigarette Smokers
Brief Title: Efficacy and Safety of Surinabant Treatment as an Aid to Smoking Cessation (SURSMOKE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6938; EUDRACT: 2006-005334-2L
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Smoking Cessation
Keywords: tobacco use cessation; cigarette smokers
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — surinabant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Active Comparator): surinabant 2,5 mg/day
  Interventions: Drug: surinabant (SR147778)
- 3 (Active Comparator): surinabant 5 mg/day
  Interventions: Drug: surinabant (SR147778)
- 4 (Active Comparator): surinabant 10 mg/day
  Interventions: Drug: surinabant (SR147778)

INTERVENTIONS:
Drug: surinabant (SR147778) — oral administration
  Arms: 2; 3; 4
Drug: placebo — oral administration
  Arms: 1

SUMMARY:
Surinabant is a new, potent and selective antagonist for the cannabinoid CB1 receptor, which might be clinically useful in the treatment of dependence to nicotine.

The primary study objective is the assessment of efficacy of 3 doses of surinabant on abstinence from smoking in cigarette smokers. The main secondary objectives are the effect of surinabant on body weight and its clinical and biological safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients over legal age smoking at least 10 cigarettes/day as a mean within the 6 months preceding the screening visit.

Exclusion Criteria:

* Patients with a limited level of motivation.
* Other participant in a household enrolled in the study.
* Patients who have smoked or consumed non-tobacco cigarettes or any form of tobacco product more than 3 days within the 3 months preceding the screening visit.
* Patients dependent to alcohol or illicit drugs.
* Patients with a diagnosis of Psychotic Disorder or currently presenting with a Depressive Episode.
* Patients who have suffered from a myocardial infarction, unstable angina or other major cardiovascular event within the past 6 months prior to screening.
* Pregnant or breast-feeding women or women not protected by effective contraceptive method of birth control.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence from tobacco smoking (including smoking diaries, measurements of carbon monoxide and cotinine) at every visit | during the last four weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in total body weight | 8 weeks
Total score of the Questionnaire of Smoking Urges | 8 weeks
Safety endpoints (physical examinations, vital signs, electrocardiograms, laboratory parameters, adverse events) | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claire VILAIN, M.D., Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Derived] Tonstad S, Aubin HJ. Efficacy of a dose range of surinabant, a cannabinoid receptor blocker, for smoking cessation: a randomized controlled clinical trial. J Psychopharmacol. 2012 Jul;26(7):1003-9. doi: 10.1177/0269881111431623. Epub 2012 Jan 4. PMID 22219220